CLINICAL TRIAL: NCT03912519
Title: Randomized Trial Comparing Parallel Versus Perpendicular Technique for Lumbar Medial Branch Radiofrequency Neurotomy
Brief Title: Parallel Versus Perpendicular Technique for Lumbar Medial Branch Radiofrequency Neurotomy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Spine Intervention Society (Unknown)
Responsible Party: Principal Investigator, Byron Schneider, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 190556
Record Dates: First submitted 2019-03-19; First posted 2019-04-11 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Back Pain Without Radiation; Low Back Pain; Lumbar Radiofrequency Neurotomy
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parallel placement of 16 gauge electrodes (Active Comparator): Parallel Group will undergo radiofrequency ablation via the approach described in Spine Intervention Practice Guidelines via 16 gauge electrodes. Specifically, the target nerve will be targeted with a parallel approach so as the electrode lay parallel to the nerves location within the sulcus formed by the neck of superior articular process and transverse process (or sacral ala for L5) cephalad to the point it is covered by the mamillo-accessory ligament.
  Interventions: Procedure: Parallel placement of 16 gauge electrodes
- Perpendicular placement with 22 gauge electrodes (Active Comparator): Perpendicular Group will undergo radiofrequency ablation via the approach described in Spine Intervention Society Practice Guidelines for medial branch blocks, using a 22 gauge electrode. Specifically, the target nerve will be targeted with a perpendicular approach so as the tip of electrode contact the nerve at some point of it course along the sulcus formed by the neck of superior articular process and transverse process (or sacral ala for L5) cephalad to the point it is covered by the mamillo-accessory ligament.
  Interventions: Procedure: Perpendicular placement with 22 gauge electrodes

INTERVENTIONS:
Procedure: Parallel placement of 16 gauge electrodes — Parallel technique
  Arms: Parallel placement of 16 gauge electrodes
Procedure: Perpendicular placement with 22 gauge electrodes — Perpendicular technique
  Arms: Perpendicular placement with 22 gauge electrodes

SUMMARY:
Low back pain is a leading cause of disability worldwide. The lumbar zygapophyseal joints (z-joints) are estimated to be the source of low back pain between 10% and 40% of the time. Observational studies have shown that lumbar medial branch radiofrequency neurotomy (LMBRFN) can be an effective treatment for z-joint low back pain. Nonetheless, other publications such as the Cochrane collaboration systematic review and the "Minimal Interventional Treatments for Participants with Chronic Low Back Pain" or "MINT" randomized controlled trial conclude that LMBRFN is not efficacious. These discrepancies in the literature may be due to differences in patient selection and procedural technique. This study aims to employ patient selection via dual medial branch block resulting in at least 80% relief on both occasions. Using this rather strict enrollment criteria, the aim of the study is to then compare LMBRFN utilizing 16 gauge needles via the "parallel" approach as endorsed by Spine Intervention Society guidelines to LMBRFN performed with 22 gauge needles and another commonly employed "perpendicular" technique similar to that approach used for medial branch blocks. The primary outcome of the study will be to determine if there is a difference in the percentage of patients with lumbar facet pain who achieve moderate or good response (improvement of Numeric Pain Rating Scale of at least 50% or 80%) or in the duration of effect (median duration of moderate or good response in those with positive outcome) between these two groups.

ELIGIBILITY:
Inclusion Criteria:

* aged > 40, capable of understanding and providing consent in English, capable of complying with the outcome instruments used, capable of attending all planned follow up visits
* unilateral or bilateral low back pain of at least 4/10 on Numeric Pain Rating Scale (NPRS) present for at least 2 months that has failed to adequately respond to at least 6 weeks of physical therapy and oral pain medication
* at least 80% improvement on two consecutive lumbar medial branch blocks of no more than a total of 4 lumbar facet joints
* beyond the above stated criteria, the decision to initiate the process of a first medial branch block is based on clinical decision making of the treating physician
* Patient consents to treatment in a shared decision-making process with the treating physician.

Exclusion Criteria:

* Those whose primary complain is lumbar radiculopathy
* Those receiving remuneration for their pain treatment (e.g., disability, worker's compensation).
* Those involved in active litigation relevant to their pain.
* Those unable to read English and complete the assessment instruments.
* Those unable to attend follow up appointments
* The patient is incarcerated.
* History of prior lumbar fusion
* Progressive motor deficit, and/or clinical signs of cauda equina or polyradiculopathy
* History of lumbar steroid injection (epidural steroid injection, sacroiliac joint steroid injection, lumbar facet steroid injection) within the prior 3 months.
* Possible pregnancy or other reason that precludes the use of fluoroscopy.
* Allergy to contrast media or local anesthetics.
* BMI>40.
* Active Systemic inflammatory arthritis (e.g., rheumatoid arthritis, ankylosing spondylitis, lupus).
* Active infection or treatment of infection with antibiotics within the past 7 days.
* Medical conditions causing significant functional disability (e.g., stroke, COPD)
* Chronic widespread pain or somatoform disorder (e.g. fibromyalgia).
* Addictive behavior, severe clinical depression, or psychotic features.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2019-08-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Clinical Outcome Measurement Brief Instrument (COMBI), Global Impression of Change | Baseline to 12 months
  Global Impression of Change; Range 0-7 0 = Very much improved 7 = Very much worse
Change in Modified Clinical Outcome Measurement Brief Instrument (COMBI), Numeric Rating Scale of Pain Intensity | Baseline to 12 months
  Numeric Rating Scale of Pain Intensity; Range 0-10 0 = No pain 10 = Pain as bad as you can imagine
Change in Modified Clinical Outcome Measurement Brief Instrument (COMBI), Pain | Baseline to 12 months
  Pain sub-scale as part of the Pain, Enjoyment, General Activity domain of COMBI; Range 0-10 0 = No Pain 10 = Pain as bad as you can image
Change in Modified Clinical Outcome Measurement Brief Instrument (COMBI), Enjoyment | Baseline to 12 months
  Enjoyment sub-scale as part of the Pain, Enjoyment, General Activity domain of COMBI; Range 0-10 0 = Does not interfere 10 = Completely interferes
Change in Modified Clinical Outcome Measurement Brief Instrument (COMBI), General Activity | Baseline to 12 months
  General Activity sub-scale as part of the Pain, Enjoyment, General Activity domain of COMBI; Range 0-10 0 = Does not interfere 10 = Completely interferes
Change in Modified Clinical Outcome Measurement Brief Instrument (COMBI), Number of Participants Not Requiring Other Healthcare | Baseline to 12 months
  Categorical Outcome; ideal would be that patients no longer require other care for the condition for which they were treated. So, the scoring is simply absolute. The instrument is neither designed nor intended for more granular analysis, on the grounds that partial reduction in doses required, but nevertheless continuation of other treatment, falls short of indicating a worthwhile, successful outcome (PubMed Identifier: 25312899).
Change in Modified Clinical Outcome Measurement Brief Instrument (COMBI), Number of Participants Returning to Work | Baseline to 12 months
  Categorical outcome; it is very relevant if return to work is achieved. Failure to return to work is too vexatious an issue, with so many determinants that it is neither efficient nor effective to bother trying to record them (Reference PMID: 25312899).
Change in Oswestry Disability Index (ODI) | Baseline to 12 months
  The questionnaire is designed to give information on how pain is affecting the ability to manage everyday life. The range of scores is 0-100%.
  0-20%: "minimal disability": The patient can cope with most living activities. Usually no treatment is indicated apart from advice on lifting sitting and exercise.
  21-40%: "moderate disability": The patient experiences more pain and difficulty with sitting, lifting and standing. Travel and social life are more difficult and they may be disabled from work. Personal care, sexual activity and sleeping are not grossly affected and the patient can usually be managed by conservative means.
  41-60%: "severe disability": Pain remains the main problem in this group but activities of daily living are affected.
  61-80%: "crippled": Back pain impinges on all aspects of the patient's life. 81-100%: These patients are either bed-bound or exaggerating their symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Byron Schneider, MD, Principal Investigator — Vanderbilt University Medical Center; Blake Fechtel, MD MSc, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No